CLINICAL TRIAL: NCT00423904
Title: Implementing Early Intervention for Alcohol Use Disorders in the General Hospital
Brief Title: Brief Alcohol Intervention in General Hospitals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: E1_P1; 01EB0120; 01EB0420
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2007-01-18 (Estimated); Status verified 2007-01

CONDITIONS: Alcohol Dependence; Alcohol Abuse; At-Risk-Drinking; Heavy Episodic Drinking
Keywords: Early intervention; Brief intervention; alcohol; general hospital
MeSH Terms: conditions — Alcoholism | interventions — Crisis Intervention

INTERVENTIONS:
Behavioral: Brief intervention

SUMMARY:
The purpose of the study is to reveal the most promising procedure for implementing alcohol screening and intervention in general hospitals and to find out, if and to which extent non-specialist health professionals can be qualified to carry out motivational intervention on their own or if there is a need for a specialized counseling services. In a randomized controlled trial, patients recruited in general hospitals and fulfilling criteria for alcohol dependence, alcohol abuse, at-risk drinking or heavy episodic drinking will be allocated to three conditions: (1) Intervention by a liaison service (LC): Counselling based on the Transtheoretical Model of behaviour change (TTM) which will be provided by staff of the study (psychologists/ social worker) trained in Motivational Interviewing (MI), (2) Intervention by hospital physicians (PC): Counselling will be provided by hospital physicians trained in MI, and (3) Control group (CC): Treatment as usual, assessment only. Outcome assessment will be conducted after 12 months and includes abstinent point prevalence rates, drinks per day, help-seeking, stage progress and cost-effectiveness analysis.

DETAILED DESCRIPTION:
Background: High prevalence rates (10 - 25 %) and a promising setting for proactive intervention strategies make the general hospital a first choice setting for secondary prevention of alcohol-related disorders. Efficient screening instruments have been developed for early detection. With regard to the severity of alcohol problem (e.g. alcohol dependence vs. heavy episodic drinking) and the motivation to change, the target group is very heterogeneous. Although there are counseling strategies that take into account this heterogeneity, there is still a lack of implementation and poor knowledge about different implementation strategies in routine care. Objectives: To evaluate the effectiveness of a proactive secondary preventive intervention based on the TTM and on MI in a representative sample of general hospital patients carried out by a liaison service versus non-specialist physicians trained in counseling techniques by staff of the study. Methods: A sample of 1,479 alcohol at-risk-drinking, alcohol abusing or alcohol dependent patients from four general hospitals detected by screening questionnaires will be assigned to (1) a group counseled by an addiction liaison service, (2) a group counseled by the physicians of the ward, and (3) to an assessment-only condition with treatment as usual. Outcome will be measured one year later and will include abstinence point prevalence rates, stage progress, help seeking, and cost-effectiveness analysis. Expected impact: The project will yield new scientific knowledge on how to implement early intervention for alcohol at-risk-drinking and alcohol use disorders in the general hospital. Results of the study shall be transferred to nationwide practice guideline proposals. The study will contribute to the improvement of the health care system as well as the education of medical students. The study is designed to reveal empirical evidence for proactive TTM-based interventions for individuals suffering from a prevalent substance use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol dependence
* Alcohol abuse
* At-risk drinking
* Heavy episodic drinking

Exclusion Criteria:

* Persons physically and mentally not capable of participating in study
* Persons with a hospital stay of less than 24 hours

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Enrollment: 1035
Dates: Start 2001-10; Study Completion 2005-08

PRIMARY OUTCOMES:
Reduced alcohol consumption
Increased alcohol-specific help-seeking

SECONDARY OUTCOMES:
Increased readiness to change drinking behaviour
Increased well-being

CONTACTS AND LOCATIONS:
Overall Officials: Jennis Freyer-Adam, Dr, Principal Investigator — University Medicine Greifswald; Ulfert Hapke, Dr, Principal Investigator — University of Applied Sciences Muenster; Ulrich John, Prof Dr, Study Director — University Medicine Greifswald

REFERENCES:
- [Background] Freyer J, Bott K, Riedel J, Wedler B, Meyer C, Rumpf HJ, John U, Hapke U. Psychometric properties of the 'Processes of Change' scale for alcohol misuse and its short form (POC-20). Addict Behav. 2006 May;31(5):821-32. doi: 10.1016/j.addbeh.2005.06.007. Epub 2005 Jul 1. PMID 15993545
- [Background] Freyer J, Coder B, Bischof G, Baumeister SE, Rumpf HJ, John U, Hapke U. Intention to utilize formal help in a sample with alcohol problems: a prospective study. Drug Alcohol Depend. 2007 Mar 16;87(2-3):210-6. doi: 10.1016/j.drugalcdep.2006.08.018. Epub 2006 Sep 18. PMID 16979304
- [Background] Freyer J, Coder B, Pockrandt C, Hartmann B, Rumpf HJ, John U, Hapke U. [General hospital patients with alcohol problems welcome counselling]. Gesundheitswesen. 2006 Jul;68(7):429-35. doi: 10.1055/s-2006-926908. German. PMID 16868869
- [Background] Freyer J, Tonigan JS, Keller S, John U, Rumpf HJ, Hapke U. Readiness to change versus readiness to seek help for alcohol problems: the development of the Treatment Readiness Tool (TReaT). J Stud Alcohol. 2004 Nov;65(6):801-9. doi: 10.15288/jsa.2004.65.801. PMID 15700519
- [Background] Freyer J, Tonigan JS, Keller S, Rumpf HJ, John U, Hapke U. Readiness for change and readiness for help-seeking: a composite assessment of client motivation. Alcohol Alcohol. 2005 Nov-Dec;40(6):540-4. doi: 10.1093/alcalc/agh195. Epub 2005 Sep 26. PMID 16186144